CLINICAL TRIAL: NCT04440826
Title: Dietary Induced Thermogenic Differences After Consumption of an Unrefined Meal, a Gluten-free Meal, and a Highly Processed Meal
Brief Title: Thermic Effect of Three Different Meals in Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1502-441
Record Dates: First submitted 2020-06-11; First posted 2020-06-22 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Weight Loss; Obesity
MeSH Terms: conditions — Weight Loss; Obesity | interventions — Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole Food Meal (Active Comparator): Whole foods meal - grilled cheese and drink meal
  Interventions: Other: Whole Food Meal
- Processed Food Meal (Experimental): Highly processed foods - grilled cheese and drink meal
  Interventions: Other: Processed Food Meal
- Gluten-Free and Lactose-Free Meal (Experimental): Gluten-free and lactose-free foods - grilled cheese and drink meal
  Interventions: Other: Gluten-free and lactose-free

INTERVENTIONS:
Other: Whole Food Meal — Whole foods meal
  Arms: Whole Food Meal
Other: Processed Food Meal — Processed food meal
  Arms: Processed Food Meal
Other: Gluten-free and lactose-free — Gluten-free and lactose-free food meal
  Arms: Gluten-Free and Lactose-Free Meal

SUMMARY:
This study will investigate the acute effect of three isocaloric meals varying in level of food processing, including a whole foods, gluten-free, and highly processed meal on energy metabolism and blood glucose in 8-12 young adult, normal weight females. A secondary aim of this proposed study is to compare palatability, satiety, and perceived energy ratings among highly processed, unrefined, and gluten-free unrefined isocaloric meals.

DETAILED DESCRIPTION:
A shift towards a diet containing large quantities of highly processed foods is believed to be a major contributor to the trends in obesity. The degree of processing of foods often affects the nutritional content of the constituents. A reduction in macromolecular complexity allows for an increased rate of digestion, meaning that the body does not have to work as hard to metabolize high processed food products. Thus, the purpose of this study is to investigate the effect on energy metabolism and blood glucose after the consumption of an unrefined, whole foods meal versus two highly processed food meals, including a common Western style meal and gluten-free meal in 8-12 young adult, normal weight females. A secondary aim of this proposed study is to compare palatability, satiety, and perceived energy ratings among highly processed, unrefined, and gluten-free unrefined isocaloric meals. It is hypothesized that an unrefined meal will induce a greater postprandial thermogenic response and a smaller blood glucose response than a highly processed or gluten-free meal. Additionally, it is hypothesized that a highly processed foods meal will be considered more palatable than an unrefined or gluten-free meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females between the ages of 18 and 24 years that have BMIs that fall in the range of 18.5 kg/m2 to 28 kg/m2.

Exclusion Criteria:

* Those with a history of celiac disease or other food allergies, metabolic disease or heart disease.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 11 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2015-05-30 (Actual); Study Completion 2015-05-30 (Actual)

PRIMARY OUTCOMES:
Thermic Effect of Meals (TEM) also known as Postprandial Thermogenesis | TEM; 45-60; 105-120; and 165-180 minutes after meal ingestion
  The total amount of calories burned after each meal will be measured using indirect calorimetry with the ventilated hood technique. Specifically, the thermic effect of each meal will be measured for a total of three hours at 45 minute intervals for 15 minutes at a time (45-60; 105-120; and 165-180 minutes)

SECONDARY OUTCOMES:
Blood Glucose Response | Baseline line 0 minutes, and 60, 120, 180 minutes postprandial
  Change in postprandial blood glucose compared baseline
Change in Hunger and Palatability Scores and Energy Level | Baseline 0 minutes, and 60, 120, 180 minutes postprandial
  Assess change in subjective hunger, fullness, satiation, palatability and energy ratings using a visual analog scale ranging from 0-100 mm
Heart Rate | Baseline 0 minutes, 60, 120, and 180 minutes postprandial
  Measure heart rate following the resting metabolic rate test
Blood Pressure | Baseline 0 minutes, 60, 120, and 180 minutes postprandial
  Measure blood pressure following the resting metabolic rate test

CONTACTS AND LOCATIONS:
Overall Officials: Mary Hoehn, MPH, Study Chair — Skidmore College

IPD SHARING:
Plan to Share IPD: No